CLINICAL TRIAL: NCT03975413
Title: Single-Arm, Non-Randomized, Time Series, Single-Subject Study: Fecal Microbiota Transplantation (FMT) in Multiple Sclerosis
Brief Title: Fecal Microbiota Transplantation (FMT) in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Professor and Director of Digestive Diseases & Nutrition, Rush University Medical Center
Other Study IDs: 18082009
Record Dates: First submitted 2019-05-28; First posted 2019-06-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: FMT; Microbiome; Gait; Longitudinal; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Fecal Collection; Fecal DNA Extraction; Blood: frozen serum, plasma & buffy coat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- N=1 MS patient: Single-Arm, Non-Randomized, Time Series, Single-Subject Study. Observational study of the FMT intervention.
  Single subject studies are based on repeated observations within an individual over time and are acknowledged as an important research method for generating scientific evidence about the health or behavior of an individual. This design is desirable when the available patient pool is limited and thus it is not optimal to randomize participants to a control arm. The subject serves as his/her own control, rather than using another individual/group.These designs are used primarily to evaluate the effect of a variety of interventions in early stage clinical research development.
  Interventions: Other: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Other: Fecal Microbiota Transplantation (FMT) — Longitudinal FMT study: Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Other Names: Taymount Clinic

SUMMARY:
Multiple sclerosis (MS) is a chronic immune central nervous system (CNS) disease of unknown cause. Recent studies suggest that gut microbiota could be a trigger for the neuro-inflammation in MS and abnormal gut microbiota composition has been reported in MS patients. These data provided scientific rationale for microbiota-directed intervention, like stool transplant, for the treatment of MS.

DETAILED DESCRIPTION:
A subject (n-of-1) clinically diagnosed with Relapsing Remitting Multiple Sclerosis (RRMS), by Rush University Neurologists, volunteered and provided written informed consent to participate in this study conducted by Rush University Medical Center's department of Digestive Diseases and Nutrition. The RRMS subject underwent a fecal microbiota transplantation (FMT) administered outside the United States, at Taymount Clinic in the Bahamas, for the treatment of their MS. Being one of the investigators' patients, the subject volunteered to donate their stool samples to the Rush University Medical Center Gastrointestinal (GI) tissue repository for microbiota interrogation at the following time points: before FMT (baseline), 3, 13, 26, 39, 52 weeks (1 year) after FMT, to determine the impact on their microbiota composition and sustainability of the change. The subject also agreed to donate their blood during the above stated time points to see if FMT affected markers of bacteria translocation and systemic inflammation. The subject also agreed to have their GI symptoms, diet, sleep, and MS related symptoms (rating scales or questionnaires), MRI (brain & spine), as well as their gait metric activity objectively assessed to see if the FMT affects these symptoms and whether any observed improvement is sustained, in this proof-of-concept study. Based on this research, the investigators hypothesize that the FMT will significantly altered the overall microbial community structure to promote the growth of short chain fatty acid (SCFA)-producing beneficial bacteria, which in turn could potentially improve the MS subject's health outcomes, neurological symptoms, and walking metrics over time. More clinical trials (larger sample size) will be needed to study the potential of FMT for the treatment of MS and to examine the long term effects. FMT is an emerging treatment approach for MS. The donor selection, the separation of fecal bacteria, the frequency of FMT, the way of infusion, the long-term safety, and efficacy are still uncertain and need to be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age.
2. Diagnosis of relapsing-remitting multiple sclerosis (RRMS) by neurology(primary specialist).
3. Presence of active lesions on brain or spinal cord MRI, in the past 1 year prior to baseline.
4. MS disease duration greater than 1 year.
5. Symptomatic (Active RRMS).
6. On MS therapy/medication greater than 4 weeks.

Exclusion Criteria:

1. Newly diagnosed multiple sclerosis.
2. Inactive relapsing-remitting multiple sclerosis (RRMS).
3. Unstable or no MS therapy/medication use.
4. Presence of symptomatically active gastrointestinal diseases such as inflammatory bowel disease or celiac disease (except for hemorrhoids, hiatal hernia, or occasional (˂3 times a week) heartburn)).
5. Pre-existent organ failure or co-morbidities as these may change GI flora: a) liver disease (cirrhosis or persistently abnormal AST or ALT that are 2X˃ normal); b) kidney disease (creatinine ˃ 2.0mg/dL); c) uncontrolled psychiatric illness; d) clinically active lung disease or decompensated heart failure; e) known HIV infection; f) alcoholism; g) transplant recipients (other than FMT); h) diabetes
6. Severe malnutrition or obesity with BMI ˃ 40.
7. Antibiotic and probiotic use (except yogurt) within 4 weeks of enrollment.
8. Chronic use of NSAIDS. A washout period of 3 weeks is needed before the subject could be enrolled into the study. Low dose aspirin is allowed.
9. Pregnant or lactating women or intention of getting pregnant during the trial period.
10. Active infection including untreated latent or active tuberculosis, HIV, hepatitis, syphilis or other major active infection.
11. Active symptomatic C. Difficile infection (colonization is not an exclusion).
12. Active gastrointestinal condition being investigated (i.e. GI bleeding, colon cancer, active GI workup); history of known or suspected toxic megacolon and/or known small bowel ileus, major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment (note that this does not include appendectomy or cholecystectomy); or history of total colectomy or bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One of the investigators' patients planned to have a fecal microbiota transplant (FMT) for treatment of their MS, at the Taymount Clinic in the Bahamas, volunteered to donate multiple sample collection time points for stool and blood. Additionally, the subject would undergo gait metric activity and MRI (brain & spine), as well as completing MS rating scales and various GI, diet and sleep clinical questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Fecal microbial community structure and functional changes over six time frames for phylum, genus and species taxonomic level bacteria, virus, fungi, and archaea. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Shotgun Metagenomics
Walking and balance changes over four time frames for stride time (seconds). | Baseline, 3 week, 13 week, 52 week
  Orthopedic gait task, side gaze gait, and alternating gaze gait metrics.
Walking and balance changes over four time frames for stride distance (meters). | Baseline, 3 week, 13 week, 52 week
  Orthopedic gait task, side gaze gait, and alternating gaze gait metrics.
Walking and balance changes over four time frames for cadence (total number of steps per minute). | Baseline, 3 week, 13 week, 52 week
  Orthopedic gait task, side gaze gait, and alternating gaze gait metrics.
Walking and balance changes over four time frames for step width (meters). | Baseline, 3 week, 13 week, 52 week
  Orthopedic gait task, side gaze gait, and alternating gaze gait metrics.
Walking and balance changes over four time frames for average pelvis forward velocity (meters per second). | Baseline, 3 week, 13 week, 52 week
  Orthopedic gait task, side gaze gait, and alternating gaze gait metrics.
Walking and balance changes over four time frames for pelvis smoothness (pelvis horizontal speed). | Baseline, 3 week, 13 week, 52 week
  Orthopedic gait task, side gaze gait, and alternating gaze gait metrics.

SECONDARY OUTCOMES:
Fecal targeted short-chain-fatty-acid metabolomics concentration changes over six time frames for acetate (mM/kg), propionate (mM/kg), butyrate (mM/kg), and total SCFA (mM/kg). | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Targeted metabolomics of short-chain-fatty-acids (SCFA).
Measurement of blood serum biomarker brain-derived neurotrophic factor (BDNF) (ng/ml) changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  ELISA (enzyme-linked immunosorbent assay)
Sleep changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Munich ChronoType Questionnaire (MCTQ). Questions about work day and free day sleep schedules, work details, and lifestyle provide data to aid in the understanding of how biological clocks work in social life, such as Roenneberg's conclusions of social jetlag. The MCTQ categorizes each participant into one of seven chronotype groups, and utilizes data on participants' midsleep phase and sleep debt to survey what "type" of sleeper each person is.
Food timing changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Food Timing Screener (FTS) questionnaire. A structured food demographics questionnaire was therefore developed to access food timing. The questionnaire consists of eight questions asking subjects' eating habits on work days and non-work days. Questions include the time of the main meal during work and non-work days, time of last meal before bed, consistency of dinner within work and non-work days, and consistency of breakfast, lunch, and dinner between work and non-work days.
Gastrointestinal symptoms changes over six time frames (t-scores, mean, standard deviations). | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Patient-Reported Outcomes Measurements Information System (PROMIS) gastrointestinal questionnaire for Belly Pain (6 questions), Bowel Incontinence (4 questions), Constipation (9 questions), and Gas & Bloating (12 questions). Higher score denoted more GI symptoms. Lower score denotes less GI symptoms. Scores range from 20 (low) to 80 (high). A score of 50 is denoted as the general population.
Walking changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Multiple sclerosis walking scale questionnaire. Higher scores indicate a greater impact from MS on walking than lower scores. Scale range from 1 (no impact) to 5 (high impact). 12 questions in total.
Lesions changes over three time frames. | Baseline, 26 week and 52 week
  MRI of brain and spine
Food and frequency of consumption changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Food Time Questionnaire (FTQ) consists of a list of foods and the frequency in which these foods are consumed in at each time frame.
Single day food recall changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Automated Self-Administered 24-Hour Recall (ASA24) Dietary Assessment. Total nutrients from all supplements reported in a given day.
Diet changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  Vioscreen Food Frequency Questionnaire (FFQ). Total of 19 measured food components collected for each time frame. Vioscreen captures comprehensive dietary behaviors in just 30 minutes. VioScreen is a unique online dietary questionnaire, management and analysis system that efficiently gathers and manages data, that immediately identify dietary "habits" and counsel for lifestyle changes.
Measurement of blood serum biomarker Interleukin-6 (IL-6) (pg/ml) changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  ELISA (enzyme-linked immunosorbent assay)
Measurement of blood serum biomarker Interleukin-* (IL-8) (pg/ml) changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  ELISA (enzyme-linked immunosorbent assay)
Measurement of blood serum biomarker Tumor necrosis factor alpha (TNFα) (pg/ml) changes over six time frames. | Baseline, 3 week, 13 week, 26 week, 39 week, 52 week
  ELISA (enzyme-linked immunosorbent assay)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarzian, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available. This pilot study of FMT in a patient with multiple sclerosis (MS) could suggest a potential effective treatment. More clinical trials (larger sample size) will be needed to study the potential of FMT for the treatment of MS and it's long term effects in the future.

REFERENCES:
- [Background] Cekanaviciute E, Yoo BB, Runia TF, Debelius JW, Singh S, Nelson CA, Kanner R, Bencosme Y, Lee YK, Hauser SL, Crabtree-Hartman E, Sand IK, Gacias M, Zhu Y, Casaccia P, Cree BAC, Knight R, Mazmanian SK, Baranzini SE. Gut bacteria from multiple sclerosis patients modulate human T cells and exacerbate symptoms in mouse models. Proc Natl Acad Sci U S A. 2017 Oct 3;114(40):10713-10718. doi: 10.1073/pnas.1711235114. Epub 2017 Sep 11. PMID 28893978
- [Background] Berer K, Gerdes LA, Cekanaviciute E, Jia X, Xiao L, Xia Z, Liu C, Klotz L, Stauffer U, Baranzini SE, Kumpfel T, Hohlfeld R, Krishnamoorthy G, Wekerle H. Gut microbiota from multiple sclerosis patients enables spontaneous autoimmune encephalomyelitis in mice. Proc Natl Acad Sci U S A. 2017 Oct 3;114(40):10719-10724. doi: 10.1073/pnas.1711233114. Epub 2017 Sep 11. PMID 28893994
- [Background] Kaskow BJ, Baecher-Allan C. Effector T Cells in Multiple Sclerosis. Cold Spring Harb Perspect Med. 2018 Apr 2;8(4):a029025. doi: 10.1101/cshperspect.a029025. PMID 29358315
- [Background] Berer K, Mues M, Koutrolos M, Rasbi ZA, Boziki M, Johner C, Wekerle H, Krishnamoorthy G. Commensal microbiota and myelin autoantigen cooperate to trigger autoimmune demyelination. Nature. 2011 Oct 26;479(7374):538-41. doi: 10.1038/nature10554. PMID 22031325
- [Background] Tremlett H, Fadrosh DW, Faruqi AA, Hart J, Roalstad S, Graves J, Lynch S, Waubant E; US Network of Pediatric MS Centers. Gut microbiota composition and relapse risk in pediatric MS: A pilot study. J Neurol Sci. 2016 Apr 15;363:153-7. doi: 10.1016/j.jns.2016.02.042. Epub 2016 Feb 20. PMID 27000242
- [Background] Ochoa-Reparaz J, Magori K, Kasper LH. The chicken or the egg dilemma: intestinal dysbiosis in multiple sclerosis. Ann Transl Med. 2017 Mar;5(6):145. doi: 10.21037/atm.2017.01.18. PMID 28462225
- [Background] Kirby TO, Ochoa-Reparaz J. The Gut Microbiome in Multiple Sclerosis: A Potential Therapeutic Avenue. Med Sci (Basel). 2018 Aug 24;6(3):69. doi: 10.3390/medsci6030069. PMID 30149548
- [Background] Adamczyk-Sowa M, Medrek A, Madej P, Michlicka W, Dobrakowski P. Does the Gut Microbiota Influence Immunity and Inflammation in Multiple Sclerosis Pathophysiology? J Immunol Res. 2017;2017:7904821. doi: 10.1155/2017/7904821. Epub 2017 Feb 20. PMID 28316999
- [Background] Camara-Lemarroy CR, Metz LM, Yong VW. Focus on the gut-brain axis: Multiple sclerosis, the intestinal barrier and the microbiome. World J Gastroenterol. 2018 Oct 7;24(37):4217-4223. doi: 10.3748/wjg.v24.i37.4217. PMID 30310254
- [Background] Makkawi S, Camara-Lemarroy C, Metz L. Fecal microbiota transplantation associated with 10 years of stability in a patient with SPMS. Neurol Neuroimmunol Neuroinflamm. 2018 Apr 3;5(4):e459. doi: 10.1212/NXI.0000000000000459. eCollection 2018 Jul. No abstract available. PMID 29619403
- [Background] Quintana FJ, Prinz M. A gut feeling about multiple sclerosis. Proc Natl Acad Sci U S A. 2017 Oct 3;114(40):10528-10529. doi: 10.1073/pnas.1714260114. Epub 2017 Sep 25. No abstract available. PMID 28973867
- [Background] Smits LP, Bouter KE, de Vos WM, Borody TJ, Nieuwdorp M. Therapeutic potential of fecal microbiota transplantation. Gastroenterology. 2013 Nov;145(5):946-53. doi: 10.1053/j.gastro.2013.08.058. Epub 2013 Sep 7. PMID 24018052
- [Background] Chu F, Shi M, Lang Y, Shen D, Jin T, Zhu J, Cui L. Gut Microbiota in Multiple Sclerosis and Experimental Autoimmune Encephalomyelitis: Current Applications and Future Perspectives. Mediators Inflamm. 2018 Apr 2;2018:8168717. doi: 10.1155/2018/8168717. eCollection 2018. PMID 29805314
- [Background] Jangi S, Gandhi R, Cox LM, Li N, von Glehn F, Yan R, Patel B, Mazzola MA, Liu S, Glanz BL, Cook S, Tankou S, Stuart F, Melo K, Nejad P, Smith K, Topcuolu BD, Holden J, Kivisakk P, Chitnis T, De Jager PL, Quintana FJ, Gerber GK, Bry L, Weiner HL. Alterations of the human gut microbiome in multiple sclerosis. Nat Commun. 2016 Jun 28;7:12015. doi: 10.1038/ncomms12015. PMID 27352007
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334